CLINICAL TRIAL: NCT03363906
Title: Relative Bioavailability of an Investigational Single Dose of Dulaglutide After Subcutaneous Administration by a Single Dose Pen Compared to a Prefilled Syringe in Healthy Subjects
Brief Title: A Study of Dulaglutide in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16878; H9X-MC-GBGM (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-12-01; First posted 2017-12-06 (Actual); Results first posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2018-07

CONDITIONS: Healthy
MeSH Terms: interventions — dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dulaglutide (Reference) (Experimental): Dulaglutide 4.5 mg administered subcutaneously (SC) in 3 prefilled syringes (PFS) in one of two study periods
  Interventions: Drug: Dulaglutide (Reference)
- Dulaglutide (Test) (Experimental): Dulaglutide 4.5 mg administered SC in 1 single dose pen (SDP) in one of two study periods
  Interventions: Drug: Dulaglutide (Test)

INTERVENTIONS:
Drug: Dulaglutide (Reference) — Administered SC
  Other Names: LY2189265
  Arms: Dulaglutide (Reference)
Drug: Dulaglutide (Test) — Administered SC
  Other Names: LY2189265
  Arms: Dulaglutide (Test)

SUMMARY:
The purpose of this study is to evaluate a new formulation of dulaglutide (study drug) administered under the skin as one injection using a single dose pen compared to three injections using a pre filled syringe.

This study will evaluate how much of the study drug enters the body and how long it takes the body to get rid of it. Information about any side effects that may occur will also be collected.

The study will last about 84 days, including screening and will require overnight stays in the clinical research unit (CRU).

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy as determined by medical history and physical examination at time of screening
* Have a body mass index of greater than or equal to (≥) 23 kilograms per meter squared (kg/m²) inclusive

Exclusion Criteria:

* Have known allergies to dulaglutide, glucagon-like peptide-1 (GLP-1) related compounds, or any components of the formulation
* Have family history of medullary thyroid cancer (MTC) or a genetic condition that predisposes to MTC
* Have a history or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis) or gastrointestinal disorder (e.g., relevant esophageal reflux or gall bladder disease) or any gastrointestinal disease which impacts gastric emptying (e.g., gastric bypass surgery, pyloric stenosis, with the exception of appendectomy) or could be aggravated by GLP-1 analogs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomly assigned into different treatment sequences. Participants in Treatment Sequence A will receive Treatment 1 then Treatment 2. Participants in Treatment Sequence B will receive Treatment 2 then Treatment 1.
Groups:
- Sequence A Dulaglutide (Reference) Then Dulaglutide (Test): Dulaglutide (4.5 milligram [mg]) administered subcutaneously (SC) in 3 prefilled syringes (PFS) in period 1 and then dulaglutide 4.5 mg administered SC in single dose pen (SDP) in period 2.
- Sequence B Dulaglutide (Test) Then Dulaglutide (Reference): Dulaglutide 4.5 mg administered SC in one (SDP) in period 1 and then Dulaglutide 4.5 mg administered SC (PFS) in period 2.
Period: Period 1 (Reference or Test)
Arm/Group | Sequence A Dulaglutide (Reference) Then Dulaglutide (Test) | Sequence B Dulaglutide (Test) Then Dulaglutide (Reference)
Started | 15 | 12
Received at Least One Dose of Study Drug | 15 | 11
Completed | 14 | 10
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 2
Period: Period 2 (Test or Reference)
Arm/Group | Sequence A Dulaglutide (Reference) Then Dulaglutide (Test) | Sequence B Dulaglutide (Test) Then Dulaglutide (Reference)
Started | 14 | 10
Received at Least One Dose of Study Drug | 12 | 9
Completed | 10 | 9
Not Completed | 4 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Dulaglutide Test and Reference: Dulaglutide 4.5 mg administered SC in 3 prefilled syringes and 1 single dose pen in one of two study periods.
Arm/Group | Dulaglutide Test and Reference
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Dulaglutide
Description: Pharmacokinetics was assessed in healthy participants to determine the area under the concentration time curve from 0 to infinity (AUC[0-∞]) of Dulaglutide.
Time Frame: Periods 1 and 2: Day 1 - 8 and Day 15: Predose, 24, 48, 72,96,120,144,168, and 336 hours post dose; Follow Up: Day 28
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data in the PFS or SDP arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram.hour/milliliter (ng.h/mL)
Groups:
- Dulaglutide (Reference): Dulaglutide 4.5 mg administered SC in 3 prefilled syringes in one of two study periods
- Dulaglutide (Test): Dulaglutide 4.5 mg administered SC in 1 single dose pen in one of two study periods
Arm/Group | Dulaglutide (Reference) | Dulaglutide (Test)
Number analyzed (Participants) | 24 | 23
nanogram.hour/milliliter (ng.h/mL) | 37400 (38) | 40000 (33)
Statistical Analysis 1: Comparison: Dulaglutide (Reference) vs Dulaglutide (Test); Test type: Superiority; p = 0.473, Mixed Models Analysis; Ratio Geometric Least Squares (LS) Mean = 1.04, 90% CI 2-sided [0.949 to 1.14]

2. Primary Outcome: PK: Maximum Observed Drug Concentration (Cmax) of Dulaglutide
Description: Pharmacokinetics was assessed in healthy participants to determine the maximum observed drug concentration (Cmax) of Dulaglutide.
Time Frame: Periods 1 and 2: Day 1 - 8 and Day 15: Predose, 24, 48, 72,96,120,144,168, and 336 hours post dose; Follow Up : Day 28
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Dulaglutide (Reference) | Dulaglutide (Test)
Number analyzed (Participants) | 24 | 23
nanogram/milliliter (ng/mL) | 213 (41) | 240 (39)
Statistical Analysis 1: Comparison: Dulaglutide (Reference) vs Dulaglutide (Test); Test type: Superiority; p = 0.119, ANOVA; Mean Difference (Final Values) = 1.14, 90% CI 2-sided [0.993 to 1.30]

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: All randomized participants who received at least one dose of study drug and had evaluable PK data in the PFS or SDP arms.
Arm/Group | Dulaglutide (Reference) | Dulaglutide (Test)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 15/24 | 14/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dulaglutide (Reference) (N=24) | Dulaglutide (Test) (N=23)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 11 (13) | 12 (15)
Vomiting (Gastrointestinal disorders) | 5 (5) | 7 (9)
Injection site pain (General disorders) | 2 (3) | 2 (2)
Dizziness (Nervous system disorders) | 4 (5) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT03363906/SAP_000.pdf
  • Study Protocol (2017-09-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT03363906/Prot_001.pdf